CLINICAL TRIAL: NCT04253483
Title: A Pilot Study Comparing High-Dose Rate Brachytherapy and Stereotactic Ablative Radiotherapy as Monotherapy in Localized Prostate Cancer
Brief Title: Comparison of High-Dose Rate Brachytherapy and Stereotactic Ablative Radiotherapy as Monotherapy for the Treatment of Localized Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lara Hathout, MD, FRCPC, Assistant Professor, Dept. of Radiation Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018002793; NCI-2020-00236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2018002793; 081805 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (HDR) (Experimental): Patients undergo HDR.
  Interventions: Radiation: High-Dose Rate Brachytherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (SABR) (Experimental): Patients undergo SABR every other day for 5 treatments.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy — Undergo HDR
  Other Names: Brachytherapy, High Dose
  Arms: Arm I (HDR)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Stereotactic Ablative Radiotherapy — Undergo SABR
  Other Names: SABR/SBRT
  Arms: Arm II (SABR)

SUMMARY:
This phase II trial compares high-dose rate brachytherapy and stereotactic ablative radiotherapy as monotherapy in treating patients with prostate cancer that has not spread to other parts of the body (localized). High-dose rate brachytherapy delivers radiation directly into the prostate within a few minutes by a single radioactive seed through temporarily placed plastic catheters inside the prostate gland. Stereotactic ablative radiotherapy is an external beam radiation method that delivers large doses of radiation to the cancer in a short period of time, usually 5 treatments. This trial aims to find which of these two approaches is better in terms of patient-reported quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess feasibility of a pilot non-randomized trial evaluating stereotactic ablative radiotherapy (SABR) and high-dose rate brachytherapy for localized prostate cancer.

OUTLINE: Patients elect to participate in arms 1 or 2.

ARM I: Patients undergo high-dose rate brachytherapy (HDR).

ARM II: Patients undergo SABR every other day for 5 treatments.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within the last 9 months. Patients on active surveillance with evidence of disease progression are eligible to the protocol as long as they meet the eligibility criteria and have a recent prostate biopsy (within 9 months)
* Low-risk and intermediate-risk patients are eligible according to the following guidelines:

  * Low and intermediate-risk disease defined as:

    * Clinical stage T1-T2 and Gleason =< 7 and prostate specific antigen (PSA) < 15 ng/ml
* Lymph node evaluation by either computed tomography (CT) or magnetic resonance imaging (MRI) and bone scan are optional and are left at the discretion of the treating physician
* Prostate MRI is recommended by not mandatory
* No alpha reductase inhibitors use within 2 weeks of randomization. A washout period of 2 weeks is required prior to randomization
* Eastern Cooperative Oncology Group status 0-1
* Judged to be medically fit for brachytherapy by a radiation oncologist
* Concurrent, neoadjuvant and/or adjuvant androgen deprivation therapy (ADT) is not permitted
* Prostate volume by trans-rectal ultrasound (TRUS) =< 60 cc
* International Prognostic Scoring System (IPSS) =< 20 (alpha blockers allowed)
* Patients must sign a study specific informed consent form prior to study entry
* Patients must by accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating center. Investigators must assure themselves that patients enrolled in this trial will be available for complete documentation of the treatment, adverse events, and follow up
* Protocol treatment is to begin within 4 weeks of patient randomization

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumors curatively treated with no evidence of disease for >= 5 years
* Prior or current bleeding diathesis
* Radical surgery for carcinoma of the prostate, prior pelvic radiation, prior chemotherapy for prostate cancer, prior transurethral resection of the prostate (TURP), prior cryosurgery of the prostate
* Stage T3b and evidence of nodal or distant metastatic disease on diagnostic CT, MRI or bone scan
* Subjects who have plans to receive other concomitant or post treatment adjuvant antineoplastic therapy while on this protocol including surgery, cryotherapy, conventionally fractionated radiotherapy, hormonal therapy, or chemotherapy given as part of the treatment of prostate cancer
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial for fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulations defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immumo-compromised patients
  * Patients with history of inflammatory colitis (including Crohn's disease and ulcerative colitis) or collagen vascular diseases including rheumatoid arthritis and lupus are not eligible
* Subjects who have a history of significant psychiatric illness
* Men of reproductive potential who do not agree that they or their partner will use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of comparing stereotactic ablative radiotherapy (SABR) and high-dose rate brachytherapy (HDRB) | 36 months
  Feasibility is defined as success in enrolling patients, performing the procedures, reporting adverse effects, collecting and managing data across several institutions and patient compliance in completing health-related quality of life questionnaires.

SECONDARY OUTCOMES:
Changes in patient reported Health-Related Quality of life (HRQoL) | Baseline up to 36 months
  Will be assessed by the Expanded Prostate Cancer Index Composite (EPIC)-26 short form at baseline, 1,3,6,9,12,18,24 and 36 months.
  The response to each EPIC item is standardized to a 0 to 100 scale, with higher scores representing better quality of life. Each domain is then scored by adding the score of each item within the group divided by the total number of items. Since androgen-deprivation therapy is not permitted in our study, the hormonal score will not be reported. HRQoL scores in the bowel, sexual, urinary incontinence and irritative domains will be evaluated.
Changes in patient-reported urinary toxicity | Baseline up to 36 months
  Will be assessed by American Urology Association Symptom Score questionnaires (AUA) at baseline, 1,3,6,9,12,18,24 and 36 months.
  The AUA evaluates urinary function, 7 questions, total score is 35. The higher the score, the higher rate of urinary toxicity.
Changes in patient-reported sexual toxicity | Baseline up to 36 months
  Will be assessed by Sexual Health Inventory for Men (SHIM) questionnaires at baseline, 1,3,6,9,12,18,24 and 36 months.
  The SHIM, score 1-25 lower score reflecting severe erectile dysfunction.
Incidence of adverse events | Baseline up to 36 months
  Physician-reported adverse events using the Common Terminology Criteria for Adverse Events version 4.0 will be reported at baseline, 1,3,6,9,12,18,24 and 36 months at each patient visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Hathout, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - RWJBarnabas Health - Saint Barnabas Medical Center, Livingston, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No